CLINICAL TRIAL: NCT03040726
Title: Fixed-Dose Netupitant and Palonosetron for Chronic Nausea and Vomiting in Cancer Patients
Brief Title: Netupitant and Palonosetron Hydrochloride in Preventing Chronic Nausea and Vomiting in Patients With Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2016-0843; NCI-2017-00599 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0843 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Results first posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Malignant Neoplasm; Nausea; Vomiting
MeSH Terms: conditions — Neoplasms; Nausea; Vomiting | interventions — netupitant; Palonosetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (netupitant, palonosetron hydrochloride) (Experimental): Patients receive netupitant orally (PO) and palonosetron hydrochloride PO on days 1, 6, and 11 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Netupitant; Drug: Palonosetron; Drug: Palonosetron Hydrochloride; Other: Questionnaire Administration
- Group II (placebo) (Placebo Comparator): Patients receive placebo PO on days 1, 6, and 11.
  Interventions: Other: Placebo; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Netupitant — Given PO
  Other Names: CID6451149; D05152; RO 67-3189/000
  Arms: Group I (netupitant, palonosetron hydrochloride)
Drug: Palonosetron — Given PO
  Arms: Group I (netupitant, palonosetron hydrochloride)
Drug: Palonosetron Hydrochloride — Given PO
  Other Names: Aloxi; RS 25259-197
  Arms: Group I (netupitant, palonosetron hydrochloride)
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Group II (placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase II/III trial studies how well netupitant and palonosetron hydrochloride works in preventing chronic nausea and vomiting in patients with cancer. Netupitant and palonosetron hydrochloride may reduce nausea and vomiting.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the efficacy (i.e. change in nausea numeric rating scale [NRS] from baseline between day 5-15) of fixed dose netupitant and palonosetron hydrochloride (palonosetron) (NEPA) for chronic nausea in cancer patients.

SECONDARY OBJECTIVES:

I. To assess the secondary outcomes (e.g. proportion of patients who achieved their personalized nausea goal, antiemetic use, nausea episodes duration/frequency) for NEPA versus (vs.) placebo.

II. To assess the adverse effects associated with NEPA and placebo.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive netupitant orally (PO) and palonosetron hydrochloride PO on days 1, 6, and 11 in the absence of disease progression or unacceptable toxicity.

GROUP II: Patients receive placebo PO on days 1, 6, and 11.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer
* Chronic nausea over the past 4 weeks
* Average nausea numeric rating scale >= 4/10 over the past 5 days at screening
* Outpatient at MD Anderson Cancer Center
* Karnofsky performance status >= 50%
* Age 18 or older
* Able to complete study assessments, including keeping a daily diary

Exclusion Criteria:

* Delirium (i.e. Memorial Delirium Rating Scale > 13)
* Clinical evidence of bowel obstruction at the time of study enrollment
* Expected to use other 5HT3 antagonists or NK1 antagonists for prophylaxis during the study
* Continuation of over-the-counter therapies for nausea and/or vomiting during the study
* On cytotoxic chemotherapy in the high/moderate/low emetogenic risk categories or oral antineoplastic agents in the high or moderate emetogenic risk categories according to the latest National Comprehensive Cancer Network (NCCN) guideline within 2 weeks of study enrollment
* On scheduled potent CYP3A4 inducers at the time of study enrollment (avasimibe, carbamazepine, phenytoin, rifampin, efavirenz, nevirapine, barbiturates, systemic glucocorticoids, modafinil, oxcarbazine, phenobarbital, pioglitazone, rifabutin, St. John's wort, troglitazone)
* On scheduled CYP3A4 substrates with narrow safety range at the time of study enrollment (alfentanil, cyclosporine, dihydroergotamine, ergotamine, pimozide, quinidine, sirolimus, tacrolimus)
* On scheduled strong or moderate CYP3A4 inhibitors (boceprevir, clarithromycin, conivaptan, indinavir, itraconazole, ketoconazole, lopinavir/ritonavir, mibefradil, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, voriconazole; amprenavir, aprepitant, atazanavir, ciprofloxacin, darunavir/ritonavir, diltiazem, erythromycin, fluconazole, fosamprenavir, grapefruit juice, imatinib, verapamil) within one week of study enrollment
* Unwilling to provide informed consent
* Severe renal impairment (calculated creatinine clearance =< 29 cc/min)

  * Calculated creatinine clearance can be done within 14 days of study enrollment
* Severe liver impairment (Child-Pugh score > 9)

  * Total (T.) bilirubin, albumin, prothrombin time, and serum creatinine tests can be done within 14 days of study enrollment (only if not performed in the last 14 days)
* Females who are pregnant, lactating, or intend to become pregnant during the participation of the study; childbearing age women who are not on birth control; positive pregnancy test for women of childbearing potential, as defined by intact uterus and ovaries, and no history of menses within the last 12 months; pregnancy test to be performed on the day of enrollment; in cases of women with elevated beta-human chorionic gonadotropin (b-HCG), these candidates will be eligible to participate so long as the level of b-HCG is not consistent with pregnancy and the non-pregnant status is confirmed by a gynecologic examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Hui D, Puac V, Shelal Z, Liu D, Maddi R, Kaseb A, Javle M, Overman M, Yennurajalingam S, Gallagher C, Bruera E. Fixed-Dose Netupitant and Palonosetron for Chronic Nausea in Cancer Patients: A Double-Blind, Placebo Run-in Pilot Randomized Clinical Trial. J Pain Symptom Manage. 2021 Aug;62(2):223-232.e1. doi: 10.1016/j.jpainsymman.2020.12.023. Epub 2021 Jan 1. PMID 33388382
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cancer patients with age >=18, chronic nausea over the past 4 weeks, an average nausea numeric rating scale (NRS) >=4/10 over the past 5 days were recruited from the Supportive Care, Gastrointestinal Medical Oncology, Breast Medical Oncology, and the Gastroenterology, Hepatology and Nutrition clinics at the University of Texas MD Anderson Cancer Center.
Pre-assignment Details: A total of 53 participants were enrolled but 46 were randomized. 7 participants were not randomized for various reasons that included "Change in cancer treatment" (n=3), "Developed renal failure" (n=1), "Developed bowel obstruction" (n=1) and "Other" (n=2)
Groups:
- Blinded Intervention gp.: Took one Netupitant/Palonosetron (NEPA) capsule every 5 days for 2 doses
- Blinded Placebo gp.: Took one Placebo capsule every 5 days for 2 doses
Period: Overall Study
Arm/Group | Blinded Intervention gp. | Blinded Placebo gp.
Started | 31 | 15
Started Placebo run-in Phase | 31 | 15
Started Blinded Phase | 22 | 11
Completed | 21 | 9
Not Completed | 10 | 6
Not completed — Reasons for not completing Placebo run in phase phase; Drop Out | 4 | 0
Not completed — Reasons for not completing Placebo run in phase phase; withdrawal | 1 | 1
Not completed — Reasons for not completing Placebo run in phase: Nausea NRS score >4 | 4 | 3
Not completed — Reasons for not completing Blinded phase: Hospitalization | 0 | 2
Not completed — Reasons for not completing Blinded phase : Withdrawal | 1 | 0

BASELINE CHARACTERISTICS:
Population: We have 2 arms in this study (intervention group and Placebo group) during randomization. These 2 arms included all participants who entered in Placebo run out phase. Baseline characteristics thus have 2 arms/groups.
Groups:
- Blinded Placebo gp.: Took Placebo capsule every 5 days for 2 doses
- Total: Total of all reporting groups
Arm/Group | Blinded Intervention gp. | Blinded Placebo gp. | Total
Number analyzed (Participants) | 31 | 15 | 46
Age, Continuous [Mean (Full Range); unit: years] | 56.2 [25 to 75] | 52.7 [27 to 69] | 55 [25 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 7 | 30
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 28 | 11 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 3 | 12
  White | 21 | 12 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 15 | 46
Cancer Stage [Count of Participants; unit: Participants]
  Metastatic | 15 | 9 | 24
  Locally advanced | 15 | 6 | 21
  Recurrent or persistent | 1 | 0 | 1
Cancer Type [Count of Participants; unit: Participants]
  Breast | 4 | 1 | 5
  Gastrointestinal | 21 | 12 | 33
  Genitourinary | 1 | 0 | 1
  Respiratory | 3 | 0 | 3
  Hematology | 1 | 0 | 1
  Gynaecological | 0 | 1 | 1
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Nausea Numerical Rating Scale (NRS) Between Day 5 and Day 15
Description: Average intensity of nausea over the past 24 hours was assessed daily using a validated numeric rating scale from 0 to 10, where 0= none and 10= worse possible nausea. The total score ranged from 0-10. We measured the within-group change in nausea intensity from day 5 to day 15. Wilcoxon rank sum test was used for analysis.
Time Frame: Day 5 and Day 15
Population: Those who completed Day 15
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Blinded Intervention Group: Netupitant/Palonosetron (NEPA) capsule every 5 days for 2 doses
- Blinded Placebo Group: Placebo capsule every 5 days for 2 doses
Arm/Group | Blinded Intervention Group | Blinded Placebo Group
Number analyzed (Participants) | 21 | 10
score on a scale | -2.0 [-3.1 to -0.8] | -2.3 [-3.9 to -0.7]
Statistical Analysis 1: Comparison: Blinded Intervention Group vs Blinded Placebo Group; Test type: Other; p = 0.98, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Functional Living Index Emesis (FLIE): Nausea Sub-score
Description: FLIE is a questionnaire validated to assess the impact of chemotherapy induced nausea and vomiting on patient's function and quality of life over the past 5 days. It consists of 18 items, with 9 items on nausea and 9 items on vomiting. Each question was rated using a Numerical Rating Scale (NRS) from 1 to 7. The total Nausea sub-score ranges from 9 to 63, where a higher score indicates higher quality of life. We measured the change of nausea sub-score between baseline 5 to day 15. Wilcoxon rank sum test was used for analysis.
Time Frame: Baseline and Day 15
Population: Those who completed Day 15
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Blinded Intervention Group. | Blinded Placebo Group
Number analyzed (Participants) | 21 | 9
score on a scale | -16.6 [-22.6 to -10.5] | -18 [-22.0 to -14.0]
Statistical Analysis 1: Comparison: Blinded Intervention Group. vs Blinded Placebo Group; Test type: Other; p = 0.40, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Functional Living Index Emesis (FLIE): Vomiting Sub-score
Description: FLIE is a questionnaire validated to assess the impact of chemotherapy induced nausea and vomiting on patient's function and quality of life over the past 5 days. It consists of 18 items, with 9 items on nausea and 9 items on vomiting. Each question was rated using a Numerical Rating Scale (NRS) from 1 to 7. The total Vomiting sub-score ranges from 9 to 63, where a higher score indicates higher quality of life. We measured the change of vomiting sub-score from baseline to day 15.Wilcoxon rank sum test was used for analysis.
Time Frame: Baseline and Day 15
Population: Those who completed Day 15
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Blinded Intervention Group | Blinded Placebo Group
Number analyzed (Participants) | 21 | 9
score on a scale | -12.5 [-20.8 to -4.2] | -9.7 [-18.2 to -1.2]
Statistical Analysis 1: Comparison: Blinded Intervention Group vs Blinded Placebo Group; Test type: Other; p = 0.79, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Index of Nausea, Vomiting and Retching: Total Experience Score
Description: Index of Nausea, Vomiting, and Retching, which consists of 8 items asking about the patient's experience regarding nausea and vomiting over the past 12 hours. Each item included a 5-point Likert scale (0-4 points) with descriptive words. Total experience score ranged from 0-32 with higher score indicates more nausea/vomiting. We measured the change in score between day 5 and day 15. Wilcoxon rank sum test was used for analysis.
Time Frame: Day 5 and Day 15
Population: Those who completed Day 15
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Blinded Intervention Group | Blinded Placebo Group
Number analyzed (Participants) | 21 | 10
score on a scale | -2.3 [-4.4 to -0.3] | -2.5 [-6.9 to 1.9]
Statistical Analysis 1: Comparison: Blinded Intervention Group vs Blinded Placebo Group; Test type: Other; p = 0.57, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Study Day 15
Description: Adverse events were assessed within 15 study days
Groups:
- Placebo gp.: Took one Placebo capsule every 5 days for 2 doses
Arm/Group | Blinded Intervention gp. | Placebo gp.
All-Cause Mortality (participants affected / at risk) | 3/30 | 2/43
Serious Adverse Events (participants affected / at risk) | 1/30 | 3/43
Other Adverse Events (participants affected / at risk) | 10/30 | 9/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blinded Intervention gp. (N=30) | Placebo gp. (N=43)
Dehydration (Gastrointestinal disorders) | 1 | 0 (0)
Hepatic failure (Gastrointestinal disorders) | 1 | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1
Acute Kidney imjury (Renal and urinary disorders) | 0 (0) | 1
Death NOS (General disorders) | 0 (0) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinded Intervention gp. (N=30) | Placebo gp. (N=43)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Edema face (General disorders) | 0 | 1
Edema legs (General disorders) | 2 | 0
Fatigue (General disorders) | 2 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT03040726/Prot_SAP_000.pdf